CLINICAL TRIAL: NCT06453447
Title: Prednisone for the Early Treatment of Complex Regional Pain Syndrome After Distal Radius Fracture - a Pilot Randomized Trial
Brief Title: Prednisone for CRPS in Distal Radius Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Principal Investigator, David Stockton, Clinical Assistant Professor, Orthopaedic Trauma Surgeon, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H23-02327
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-06

CONDITIONS: Complex Regional Pain Syndromes; Distal Radius Fractures
Keywords: wrist fracture; pain; orthopaedic surgery
MeSH Terms: conditions — Complex Regional Pain Syndromes; Wrist Fractures; Pain | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone (Experimental): 40 mg PO once daily for 14 days starting day of surgery
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): placebo tablet PO once daily for 14 days starting day of surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — 40 mg PO once daily for 14 days starting day of surgery
  Arms: Prednisone
Drug: Placebo — Placebo tablet (cellulose) PO once daily for 14 days starting day of surgery
  Arms: Placebo

SUMMARY:
Wrist fractures are the most prevalent adult fracture. Complex regional pain syndrome (CRPS) is a common complication that can occur, leading to permanent disability and is costly to the patient and healthcare system. In addition, amidst the opioid epidemic, the risk of increased opioid use in patients with CRPS prompts the need to find viable treatment strategies. This study aims to evaluate an anti-inflammatory medication, prednisone, in the early treatment of CRPS. Patients with wrist fractures who undergo surgical treatment will be randomized to receiving placebo vs prednisone for 2 weeks. Clinical assessments in the follow up period will be compared.

DETAILED DESCRIPTION:
Purpose:

Distal radius fractures are the most prevalent adult fracture, accounting for 17.5% of all fractures. Complex regional pain syndrome (CRPS) is a common complication that can occur in this population, with a reported incidence of up to 32%. CRPS can lead to permanent disability and is costly to the patient and to the healthcare system, with an estimated cumulative outpatient and pain prescription cost of $42,026 over 8 years after diagnosis. In addition, amidst the opioid epidemic, the risk of increased opioid use in patients with CRPS prompts the need to find viable treatment strategies.

While there have been various proposed treatment modalities, evidence from randomized studies is lacking. Several small studies (retrospective and prospective case series) have shown potential efficacy of glucocorticoids for the treatment of CRPS. To our knowledge, there are no randomized controlled trials that evaluate treatment of CRPS in distal radius fractures with glucocorticoids.

The purpose of this pilot study is to evaluate a short course of oral prednisone as potential treatment for patients identified as developing early signs of CRPS after sustaining a distal radius fracture that was treated operatively. We will examine feasibility metrics including patient recruitment rate, adherence to allocation and protocol, withdrawal from study, and follow-through, in order to inform design of a definitive clinical trial. We will also assess the resolution of CRPS, post-operative opioid use, and any adverse events in patients who sustain a distal radius fracture after receiving prednisone vs placebo for 2 weeks post-operatively, with 6 months follow up post injury.

Hypothesis:

We hypothesize that the proposed pilot trial will demonstrate feasibility of a future definitive trial.

In addition, we hypothesize that there will be higher rates of CRPS resolution, lower amounts of opioid consumption, and no increased adverse effects, and better clinical outcomes in patients who receive prednisone treatment compared to those who received placebo. However, formal hypothesis testing will not be performed for this pilot trial.

Justification:

Developing CRPS after sustaining a distal radius fracture can lead to devastating outcomes, including permanent disability, opioid dependency, and the inability to return to work. In addition, diagnosing CRPS can be a prolonged process due to the range of vague symptoms on presentation, which can lead to delay in treatment and worsening of outcomes. Patients with CRPS may require more follow-up and referrals, which further burdens the healthcare system.

The pathogenesis of CRPS is complex and not fully known; evidence suggests nervous system sensitisation, autonomic dysfunction, and inflammatory changes. There are numerous treatment options for CRPS, though little high-quality evidence supports their efficacy. These include but are not limited to oral anti-depressants, parenteral lidocaine and corticosteroids, surgical treatment with compressed nerve release, counselling, and occupational and physical therapy. Vitamin C has been proposed as effective prophylaxis for CRPS in distal radius fractures but data have been conflicting, with the most recent randomized controlled trial (RCT) in 2014 by Ekrol et al. showing no difference in functional outcomes or rate of CRPS in patients with distal radius fractures given Vitamin C versus placebo.

Given the prevalence of distal radius fractures in adults, a relatively high CRPS incidence in this population, and no established efficacious treatment options, more research is needed to determine evidence-based and effective treatment options for this destructive condition. Studies have identified that using glucocorticoids can potentially be effective and safe for treating patients with CRPS, possibly due to the anti-inflammatory properties of glucocorticoids. One retrospective study of patients undergoing surgery for terrible triad elbow (complex elbow fracture dislocation) injuries demonstrated improved elbow range of motion for patients receiving intraoperative dexamethasone and 6-day oral course of methylprednisolone compared to patients who did not, with no increased postoperative infection. Furthermore, the anti-inflammatory nature of glucocorticoids deserves investigation for its potential to decrease opioid consumption after distal radius surgery.

A variety of doses and duration of glucocorticoids have been used in studies to manage CRPS, with a recent review article by Kwak et al showing starting doses between 30 mg to 100 mg of prednisolone. Although glucocorticoids are known to be associated with adverse effects, most are only seen with long term therapy. In addition, studies have shown that a short-course of glucocorticoids (less than 3 to 4 weeks), irrespective of dose, do not require a tapering regimen and is not associated with increased risk of adrenal insufficiency. While osteoporosis and fracture non-union are known adverse events of long-term glucocorticoid use, this has not been demonstrated in literature for short-term use. Moreover, given the risk of non-union in distal radius fractures is exceedingly rare (0.2%), this calls for less concern for using glucocorticoids in this population.

Therefore, evaluating prednisone, a relatively cheap, accessible, and safe oral medication when used for a short duration, as an anti-inflammatory and potential early treatment agent for CRPS in distal radius fractures in this pilot study may have implications for the complication profile and functional outcome for this common fracture.

Research Design:

This will be a pilot double-blind randomized control trial in patients who sustain a distal radius fracture treated operatively with a volar locked plate and identified as at risk of developing CRPS. Follow up will be 6 months, involving 4 study visits that correspond to standard post-operative clinic visits.

Statistical Analysis:

A power analysis assuming incidence of 20% CRPS and absolute risk reduction (ARR) of 10% with prophylaxis yielded a sample size of 199 patients per arm, with 80% power and significance level (α) of 0.05 (performed using online sample size calculator at clincalc.com/stats/samplesize.aspx). Incidence and ARR were estimated based on previous RCTs assessing Vitamin C as prophylaxis for CRPS in distal radius fractures. We aim to recruit 10% for this pilot study, with 20 per arm (placebo vs prednisone), for a total of 40 patients.

The CONSORT guidelines for reporting of randomized pilot and feasibility trial will be followed for the analysis and reporting of results. An intention-to-treat analysis will be utilized.

Primary Outcomes: Descriptive statistics, reported as count and percentage, will be used to summarize the feasibility outcomes (95% CI). Table 2 presents the traffic lights criteria for each outcome of the pilot study. Green indicates feasible, red indicates not feasible, and yellow indicates likely feasible but will require adjustments to the protocol. (please see attached protocol)

Secondary and Tertiary Outcomes: Chi-square (or Fisher's Exact) test will be used to compare the proportion of CRPS between groups. Either Mann-Whitney U test or two-sample t test will be used for the other quantitative outcomes depending on the variable distribution. Multivariable regression analysis will be conducted to test for associations between the intervention and each outcome, controlling for differences in patient characteristics. All P values will be 2-sided and statistical significance will be set at P < 0.05. For this pilot trial, formal hypothesis testing will not be performed as it is underpowered.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 19 years or older;
2. Patient has a unilateral, closed, distal radius fracture confirmed by radiographs;
3. The fracture is acute, within 14 days of injury;
4. Patient undergoes open reduction internal fixation with volar locking plate;
5. Patient is identified as at risk of developing CRPS with 2 or more of the following:

   1. Pain score on visual analogue scale (VAS) greater than or equal to 5/10 within 1 week of injury and beyond;
   2. Centre of Epidemiologic Studies Depression (CES-D) score on presentation is greater than or equal to 16;
   3. Patient identifies as female;
6. Patient is identified as developing signs of CRPS based on the Budapest CRPS Criteria;
7. Patient provides informed consent.

Exclusion Criteria:

1. Patient has previously fractured ipsilateral wrist;
2. Patient has neurovascular injury associated with distal radius fracture;
3. Patient has associated extremity or polytrauma injuries that would interfere with rehabilitation and outcome measurements, in the opinion of the investigator;
4. Patient has allergy to prednisone or placebo ingredients;
5. Patient has contraindication to prednisone or placebo ingredients;
6. Patient already takes a glucocorticoid medication;
7. Patient has active bacterial, viral, or fungal infection;
8. Patient is diagnosed with diabetes;
9. Patient is pregnant, planning on becoming pregnant, or breastfeeding;
10. Patient is anticipated to have difficulty completing study follow up, in the opinion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient recruitment | 6 months
  Percentage of patients approached for recruitment who consent to study participation
Proportion of patient adherence to treatment allocation and protocol - determined by patient self-reporting | 6 months
  Percentage of patients enrolled in the study who report to completing their 14-day course of treatment
Proportion of patients with missing data from secondary and tertiary outcomes | 6 months
  Percentage of enrolled patients who do not have complete secondary and tertiary outcome measures
Proportion of patient consent withdrawal from the study | 6 months
  Percentage of patients enrolled in the study who withdraw before completion of the study
Proportion of complete patient follow up at 6 months | 6 months
  Percentage of enrolled patients who complete all follow up visits

SECONDARY OUTCOMES:
Resolution of CRPS | 2 weeks, 6 weeks, 3 months, 6 months
  The treating surgeon or care team will determine whether patients continue to meet criteria for CRPS diagnosis based on the Budapest CRPS Criteria
Total opioid consumption | 2 weeks
  Total opioids consumed post-op converted to morphine milligram equivalents by assessing remaining hydromorphone tablets
Adverse effects | 2 weeks, 6 weeks, 3 months, 6 months
  Adverse effects will be recorded. These can include but are not limited to mood changes, altered sleep, swelling of extremities, dizziness, headache, weight gain, elevated blood glucose, elevated blood pressure, upset stomach, gastrointestinal bleeding, wound complications, myopathy, infections, venous thromboembolism, hear failure, and adrenal insufficiency.

OTHER OUTCOMES:
Visual analogue scale (VAS) pain score | 2 weeks, 6 weeks, 3 months, 6 months
  Score out of 10 to monitor pain level
Centre of Epidemiologic Studies Depression (CES-D) score | 2 weeks, 6 weeks, 3 months, 6 months
  to monitor for presence of depression
Short Form-36 item (SF-36) questionnaire | 2 weeks, 6 weeks, 3 months, 6 months
  to measure patient reported quality of life
Passive wrist range of motion (ROM) | 2 weeks, 6 weeks, 3 months, 6 months
  dorsiflexion, palmarflexion, supination, pronation, and finger to palm distance will be measured and recorded by the physiotherapist at each follow up visit
The disabilities of the arm, shoulder, and hand (DASH) questionnaire | 2 weeks, 6 weeks, 3 months, 6 months
  to measure patient reported upper extremity disability and symptoms
The Brief Resiliency Scale (BRS) questionnaire | 2 weeks, 6 weeks, 3 months, 6 months
  to assess patient reported ability to cope with stress

CONTACTS AND LOCATIONS:
Overall Officials: David Stockton, MD, MASc, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Background] Moseley GL, Herbert RD, Parsons T, Lucas S, Van Hilten JJ, Marinus J. Intense pain soon after wrist fracture strongly predicts who will develop complex regional pain syndrome: prospective cohort study. J Pain. 2014 Jan;15(1):16-23. doi: 10.1016/j.jpain.2013.08.009. Epub 2013 Nov 19. PMID 24268113
- [Background] Jo YH, Kim K, Lee BG, Kim JH, Lee CH, Lee KH. Incidence of and Risk Factors for Complex Regional Pain Syndrome Type 1 after Surgery for Distal Radius Fractures: A Population-based Study. Sci Rep. 2019 Mar 19;9(1):4871. doi: 10.1038/s41598-019-41152-x. PMID 30890732
- [Background] Jellad A, Salah S, Ben Salah Frih Z. Complex regional pain syndrome type I: incidence and risk factors in patients with fracture of the distal radius. Arch Phys Med Rehabil. 2014 Mar;95(3):487-92. doi: 10.1016/j.apmr.2013.09.012. Epub 2013 Sep 29. PMID 24080349
- [Background] Elsamadicy AA, Yang S, Sergesketter AR, Ashraf B, Charalambous L, Kemeny H, Ejikeme T, Ren X, Pagadala P, Parente B, Xie J, Lad SP. Prevalence and Cost Analysis of Complex Regional Pain Syndrome (CRPS): A Role for Neuromodulation. Neuromodulation. 2018 Jul;21(5):423-430. doi: 10.1111/ner.12691. Epub 2017 Sep 29. PMID 28961359
- [Background] Kowalski C, Ridenour R, McNutt S, Ba D, Liu G, Bible J, Aynardi M, Garner M, Leslie D, Dhawan A. Risk Factors For Prolonged Opioid Use After Spine Surgery. Global Spine J. 2023 Apr;13(3):683-688. doi: 10.1177/21925682211003854. Epub 2021 Apr 15. PMID 33853404
- [Background] Atalay NS, Ercidogan O, Akkaya N, Sahin F. Prednisolone in complex regional pain syndrome. Pain Physician. 2014 Mar-Apr;17(2):179-85. PMID 24658479
- [Background] Bianchi C, Rossi S, Turi S, Brambilla A, Felisari G, Mascheri D. Long-term functional outcome measures in corticosteroid-treated complex regional pain syndrome. Eura Medicophys. 2006 Jun;42(2):103-11. PMID 16767061
- [Background] Winston P. Early Treatment of Acute Complex Regional Pain Syndrome after Fracture or Injury with Prednisone: Why Is There a Failure to Treat? A Case Series. Pain Res Manag. 2016;2016:7019196. doi: 10.1155/2016/7019196. Epub 2016 Apr 30. PMID 27445622
- [Background] Jamroz A, Berger M, Winston P. Prednisone for Acute Complex Regional Pain Syndrome: A Retrospective Cohort Study. Pain Res Manag. 2020 Feb 25;2020:8182569. doi: 10.1155/2020/8182569. eCollection 2020. PMID 32184912
- [Background] Desai MJ, Matson AP, Ruch DS, Leversedge FJ, Aldridge JM 3rd, Richard MJ. Perioperative Glucocorticoid Administration Improves Elbow Motion in Terrible Triad Injuries. J Hand Surg Am. 2017 Jan;42(1):41-46. doi: 10.1016/j.jhsa.2016.11.011. PMID 28052827
- [Background] Dutton LK, Rhee PC. Complex Regional Pain Syndrome and Distal Radius Fracture: Etiology, Diagnosis, and Treatment. Hand Clin. 2021 May;37(2):315-322. doi: 10.1016/j.hcl.2021.02.013. PMID 33892884
- [Background] Shim H, Rose J, Halle S, Shekane P. Complex regional pain syndrome: a narrative review for the practising clinician. Br J Anaesth. 2019 Aug;123(2):e424-e433. doi: 10.1016/j.bja.2019.03.030. Epub 2019 May 2. PMID 31056241
- [Background] Li Z, Smith BP, Tuohy C, Smith TL, Andrew Koman L. Complex regional pain syndrome after hand surgery. Hand Clin. 2010 May;26(2):281-9. doi: 10.1016/j.hcl.2009.11.001. PMID 20494753
- [Background] Jupiter JB, Seiler JG 3rd, Zienowicz R. Sympathetic maintained pain (causalgia) associated with a demonstrable peripheral-nerve lesion. Operative treatment. J Bone Joint Surg Am. 1994 Sep;76(9):1376-84. doi: 10.2106/00004623-199409000-00013. PMID 8077268
- [Background] Zollinger PE, Tuinebreijer WE, Kreis RW, Breederveld RS. Effect of vitamin C on frequency of reflex sympathetic dystrophy in wrist fractures: a randomised trial. Lancet. 1999 Dec 11;354(9195):2025-8. doi: 10.1016/S0140-6736(99)03059-7. PMID 10636366
- [Background] Zollinger PE, Tuinebreijer WE, Breederveld RS, Kreis RW. Can vitamin C prevent complex regional pain syndrome in patients with wrist fractures? A randomized, controlled, multicenter dose-response study. J Bone Joint Surg Am. 2007 Jul;89(7):1424-31. doi: 10.2106/JBJS.F.01147. PMID 17606778
- [Background] Ekrol I, Duckworth AD, Ralston SH, Court-Brown CM, McQueen MM. The influence of vitamin C on the outcome of distal radial fractures: a double-blind, randomized controlled trial. J Bone Joint Surg Am. 2014 Sep 3;96(17):1451-9. doi: 10.2106/JBJS.M.00268. PMID 25187584
- [Background] Kwak SG, Choo YJ, Chang MC. Effectiveness of prednisolone in complex regional pain syndrome treatment: A systematic narrative review. Pain Pract. 2022 Mar;22(3):381-390. doi: 10.1111/papr.13090. Epub 2021 Nov 25. PMID 34779145
- [Background] Beuschlein F, Else T, Bancos I, Hahner S, Hamidi O, van Hulsteijn L, Husebye ES, Karavitaki N, Prete A, Vaidya A, Yedinak C, Dekkers OM. European Society of Endocrinology and Endocrine Society Joint Clinical Guideline: Diagnosis and therapy of glucocorticoid-induced adrenal insufficiency. Eur J Endocrinol. 2024 May 2;190(5):G25-G51. doi: 10.1093/ejendo/lvae029. PMID 38714321
- [Background] Henzen C, Suter A, Lerch E, Urbinelli R, Schorno XH, Briner VA. Suppression and recovery of adrenal response after short-term, high-dose glucocorticoid treatment. Lancet. 2000 Feb 12;355(9203):542-5. doi: 10.1016/S0140-6736(99)06290-X. PMID 10683005
- [Background] Aslan M, Simsek G, Yildirim U. Effects of short-term treatment with systemic prednisone on bone healing: an experimental study in rats. Dent Traumatol. 2005 Aug;21(4):222-5. doi: 10.1111/j.1600-9657.2005.00300.x. PMID 16026529
- [Background] Prommersberger KJ, Fernandez DL. Nonunion of distal radius fractures. Clin Orthop Relat Res. 2004 Feb;(419):51-6. doi: 10.1097/00003086-200402000-00009. PMID 15021131
- [Background] Yeoh JC, Pike JM, Slobogean GP, O'Brien PJ, Broekhuyse HM, Lefaivre KA. Role of Depression in Outcomes of Low-Energy Distal Radius Fractures in Patients Older Than 55 Years. J Orthop Trauma. 2016 May;30(5):228-33. doi: 10.1097/BOT.0000000000000514. PMID 27101161
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Atkins RM, Duckworth T, Kanis JA. Features of algodystrophy after Colles' fracture. J Bone Joint Surg Br. 1990 Jan;72(1):105-10. doi: 10.1302/0301-620X.72B1.2298766.